CLINICAL TRIAL: NCT02448264
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of BCX7353 in Healthy Subjects
Brief Title: First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BCX7353 in Healthy Western and Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCX7353-101
Record Dates: First submitted 2015-05-13; First posted 2015-05-19 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Hereditary Angioedema
Keywords: kallikrein inhibitor; oral prophylaxis; BioCryst; first-in-human; hereditary angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — berotralstat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCX7353 (Experimental): BCX7353 capsules administered orally
  Interventions: Drug: BCX7353
- Placebo (Placebo Comparator): Placebo to Match BCX7353 capsules, administered orally
  Interventions: Drug: Placebo to match BCX7353

INTERVENTIONS:
Drug: BCX7353
  Arms: BCX7353
Drug: Placebo to match BCX7353
  Arms: Placebo

SUMMARY:
This is a 3-part Phase 1 dose-ranging study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single (Part 1) and multiple (Part 2) ascending doses of BCX7353 in healthy subjects, and single and multiple doses of BCX7353 in healthy Japanese subjects. Pharmacokinetics is an analysis of how the body handles the study drug BCX7353 and pharmacodynamics is an analysis of the activity the study drug BCX7353 may have in the body.

DETAILED DESCRIPTION:
Up to 6 ascending, single dose cohorts are planned to be dosed in a sequential manner in Part 1 of the study. Eight subjects will be treated with a single dose of study drug per dose cohort (6 subjects per cohort will receive BCX7353 and 2 subjects per cohort will receive matching placebo). Escalation to the next higher dose level will occur only after completion of a review of clinical safety and pharmacokinetics by the Sponsor and PI.

Up to 4 ascending, multiple dose cohorts will be enrolled in a sequential manner in Part 2 of the study. Twelve subjects will be treated with study drug per dose cohort (10 subjects will receive BCX7353 and 2 subjects will receive placebo per cohort). The planned doses, dosing regimens, and duration of dosing (7 or 14 days) for each of the Part 2 cohorts will be determined based upon safety and pharmacokinetic data collected during the study. Escalation to the next higher dose level in Part 2 will occur only after completion of a review of clinical safety and pharmacokinetics by the Sponsor and clinical site study physician.

In Part 3 of the study, the safety, tolerability, PK, and PD of single and multiple doses of oral BCX7353 versus placebo in healthy subjects of Japanese origin will be evaluated. In the single dose cohort, 16 Japanese subjects will be randomized into a single cohort to receive either placebo or 1 of 2 active doses of BCX7353. In the multiple dose cohort, twelve subjects will be treated with study drug (10 subjects will receive BCX7353 and 2 subjects will receive placebo per cohort). The planned doses (single and multiple dose cohort), and dosing regimen and duration of dosing (7 or 14 days; multple dose cohort) for Part 3 will be determined based upon safety and pharmacokinetic data collected during Parts 1 and 2 of the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent
* Body mass index 19 to 32 kg/m2 and a weight of at least 50 kg
* Abides by study restrictions
* Attends all study visits and agrees to remain in study center for the confinement period
* Acceptable birth control measures for male subjects and women of childbearing potential
* Part 3 only: Japanese subjects enrolled in Part 3 must be first generation: born in Japan, not having lived outside Japan > 5 years, able to trace maternal and paternal Japanese ancestry, with no significant change in lifestyle, including diet (at least one Japanese meal consumed per day), since leaving Japan.

Key Exclusion Criteria:

* Clinically significant medical history, current medical or psychiatric condition. This includes a history of clinically significant gastrointestinal, hematologic, renal, hepatic, bronchopulmonary, neurological, or cardiac disease
* Clinically significant ECG finding, vital sign measurement or laboratory/urinalysis abnormality at screening or baseline
* Use of over the counter medication within 7 days of dosing and anticipated use through the follow-up visit
* Use of prescription medication within 14 days of dosing and anticipated use through the follow-up visit
* Participation in any other investigational drug study within 90 days of screening
* Recent or current history of alcohol or drug abuse
* Regular recent use of tobacco or nicotine products
* Positive serology for HBV, HCV, or HIV
* Pregnant or nursing
* Donation or loss of greater than 400 mL of blood within 3 months
* Serious adverse reaction or serious hypersensitivity to any drug

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adverse events | Part 1 and Part 3 single dose cohort: absolute and change from baseline through Study Day 7; Part 2 and Part 3 multiple dose cohort: absolute and change from baseline through 14 or 21 days (depending on dosing duration)
Laboratory analyses | Part 1 and Part 3 single dose cohort: absolute and change from baseline through Study Day 7; Part 2 and Part 3 multiple dose cohort: absolute and change from baseline through 14 or 21 days (depending on dosing duration)
Vital signs | Part 1 and Part 3 single dose cohort: absolute and change from baseline through Study Day 7; Part 2 and Part 3 multiple dose cohort: absolute and change from baseline through 14 or 21 days (depending on dosing duration)
Electrocardiograms | Part 1 and Part 3 single dose cohort: absolute and change from baseline through Study Day 7; Part 2 and Part 3 multiple dose cohort: absolute and change from baseline through 14 or 21 days (depending on dosing duration)
Physical examination findings | Part 1 and Part 3 single dose cohort: absolute and change from baseline through Study Day 7; Part 2 and Part 3 multiple dose cohort: absolute and change from baseline through 14 or 21 days (depending on dosing duration)

SECONDARY OUTCOMES:
Plasma BCX7353 Cmax | plasma pharmacokinetic parameters are based on blood sampling through Day 5 for Part 1 and Part 3 single dose cohort and through Day 14 or 21 for Part 2 and Part 3 multiple dose cohort (Day depends on dosing duration)
Plasma BCX7353 Tmax | plasma pharmacokinetic parameters are based on blood sampling through Day 5 for Part 1 and Part 3 single dose cohort and through Day 14 or 21 for Part 2 and Part 3 multiple dose cohort (Day depends on dosing duration)
Plasma BCX7353 average steady-state concentration | steady-state plasma pharmacokinetic parameters are based on blood sampling through Day 14 or 21 for Part 2 and Part 3 multiple dose cohort (Day depends on dosing duration)
Plasma BCX7353 AUCinf | plasma pharmacokinetic parameters are based on blood sampling through Day 5 for Part 1 and Part 3 single dose cohort
Plasma BCX7353 AUCtau | steady-state plasma pharmacokinetic parameters are based on blood sampling through Day 14 or 21 for Part 2 and Part 3 multiple dose cohort (Day depends on dosing duration)
Plasma BCX7353 AUC0-t | plasma pharmacokinetic parameters are based on blood sampling through Day 5 for Part 1 and Part 3 single dose cohort and through Day 14 or 21 for Part 2 and Part 3 multiple dose cohort (Day depends on dosing duration)
Plasma BCX7353 t1/2 | plasma pharmacokinetic parameters are based on blood sampling through Day 5 for Part 1 and Part 3 single dose cohort and through Day 14 or 21 for Part 2 and Part 3 multiple dose cohort (Day depends on dosing duration)
Plasma BCX7353 apparent oral clearance | plasma pharmacokinetic parameters are based on blood sampling through Day 5 for Part 1 and Part 3 single dose cohort and through Day 14 or 21 for Part 2 and Part 3 multiple dose cohort (Day depends on dosing duration)
Plasma BCX7353 apparent volume of distribution | plasma pharmacokinetic parameters are based on blood sampling through Day 5 for Part 1 and Part 3 single dose cohort and through Day 14 or 21 for Part 2 and Part 3 multiple dose cohort (Day depends on dosing duration)
Plasma BCX7353 accumulation ratio | steady-state plasma pharmacokinetic parameters are based on blood sampling through Day 14 or 21 for Part 2 and Part 3 multiple dose cohort (Day depends on dosing duration)
Plasma pharmacodynamics of BCX7353 | plasma pharmacokinetic parameters are based on blood sampling through Day 5 for Part 1 and Part 3 single dose cohort and through Day 14 or 21 for Part 2 and Part 3 multiple dose cohort (Day depends on dosing duration)
  Outcome evaluated by change from baseline in ex vivo kallikrein inhibition

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Collier, MBChB, FFPM, Dip Stats (OU), Principal Investigator — Quotient Clinical Ltd
Locations (1):
- Quotient Clinical, Ruddington, United Kingdom